CLINICAL TRIAL: NCT06140121
Title: Immersive Technology to Improve Physical Therapy Engagement
Acronym: iMOVE-G
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 72980
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Physical Health
Keywords: Virtual Reality; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: VRPT then Traditional PT (Experimental): Participants will receive Virtual Reality assisted Physical Therapy sessions (VRPT) in the first Physical Therapy (PT) session and will receive traditional Physical Therapy sessions (standard care) in the second Physical Therapy session under the supervision of the accredited physical therapist.
  Interventions: Behavioral: Virtual Reality Physical Therapy; Behavioral: Traditional Physical Therapy
- Traditional PT then VRPT (Experimental): Participants will receive traditional Physical Therapy (PT) sessions (standard care) in the first Physical Therapy session and receive Virtual Reality assisted Physical Therapy sessions (VRPT) in the second Physical Therapy session under the supervision of the accredited physical therapist.
  Interventions: Behavioral: Virtual Reality Physical Therapy; Behavioral: Traditional Physical Therapy

INTERVENTIONS:
Behavioral: Virtual Reality Physical Therapy — Participants are allowed to freely choose one game from the game list. Participant will be asked to wear a validated activity tracker - ActiGraph. Baseline heart rate will be collected for 1 minute. Participants will be wearing the ActiGraph during Physical Therapy session. Participants receiving VR intervention will be instructed to wear an Oculus Quest 2 headset (Meta, Inc., Menlo Park, CA) and participate in VR applications under the supervision of the physical therapist.
  Other Names: VRPT
Behavioral: Traditional Physical Therapy — Participants will receive traditional Physical Therapy sessions (standard care) under the supervision of the accredited physical therapist. Participants will be wearing the Actigraph during Physical Therapy session. Participants will perform regular physical exercise, such as 20 minutes walking or biking on a stationary bike, under the supervision of a physical therapist.

SUMMARY:
This is an experimental study to evaluate the efficacy of a Virtual Reality aid Physical Therapy (VRPT) in increasing the physical activity levels and quality of life of children.

ELIGIBILITY:
Inclusion Criteria:

* Between age 7-25
* has an active physical therapy consultation
* Anticipated inpatient stay for more than 2 days

Exclusion Criteria:

* Legal guardian not present to obtain consent
* child with a significant neurological condition, or major developmental disability
* child with active infection of the face or hand
* a history of severe motion sickness
* a history of seizures cause by flashing light
* Major surgery within the last 48 hours

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
ActiGraph data points | During physical therapy session
  Compare the total Metabolic Equivalent of Task (METs) rate of pediatric patients when undergo virtual reality assisted physical therapy and traditional physical therapy measured by ActiGraph watch

SECONDARY OUTCOMES:
Total movement with wearable movement sensor | During physical therapy session
  Compare the total movement of pediatric patients when undergo virtual reality assisted physical therapy and traditional physical therapy measured by ActiGraph watch
Perceived exertion | baseline, during physical therapy session, immediately after the physical therapy session
  Patients will self-report perceived exertion according to the Adult OMNI-Walk/Run RPE Scale (OMNI RPE) scale after both the VR and standard of care portion. The OMNI RPE is an 11-categories perceived exertion rating scale with a numerical rating from 0 to 10 (0= Not Tired at All, 10= Very, Very Tired).
Difference in Fatigue - Short Form 10a questionnaire result | immediately after the physical therapy session
  Measured by comparison PROMIS Pediatric Item Bank GenPop v2.0 - Fatigue - Short Form 10a of patient in first physical therapy session and second physical therapy session .
  PROMIS Pediatric Item Bank GenPop v3.0 - Fatigue - Short Form 10a is a 10 items -questionnaire which measures the fatigue scale of the patient with scores range from 1 to 5,(1 = never and 5 = Almost always).
Change in current mental well being as measured by the modified WHO (Five) Well-Being Index | immediately after the physical therapy session
  The modified WHO (Five) Well-Being Index is a participant-reported outcome measure that assesses current mental well being. Questionnaire contains 5 questions . Scores range from 0 to 5, with higher scores indicating the corresponding feeling exists all the time
Acceptability of Intervention Measure (AIM) | immediately after the physical therapy session
  Acceptability, of the traditional physical therapy or virtual reality physical therapy interventions will be assessed using the Acceptability of Intervention Measure (AIM) which is a subscale of the Triple P Tool. Scale items are scored on a Likert scale from 1 to 5 where higher scores indicate higher acceptability of the intervention.
Intervention Appropriateness Measure (IAM) | immediately after the physical therapy session
  Appropriateness, of the traditional physical therapy or virtual reality physical therapy interventions will be assessed using the Intervention Appropriateness Measure (IAM) which is a subscale of the Triple P Tool. Scale items are scored on a Likert scale from 1 to 5 where higher scores indicate higher appropriateness of the intervention.
Feasibility of Intervention Measure (FIM) | immediately after the physical therapy session
  Feasibility, of the traditional physical therapy or virtual reality physical therapy interventions will be assessed using the Feasibility of Intervention Measure (FIM) which is a subscale of The Triple P Tool. Scale items are scored on a Likert scale from 1 to 5 where higher scores indicate higher feasibility.
Feasibility and acceptability survey(patient) | immediately after the physical therapy session
  This is an self developed feasibility survey. Feasibility, of the virtual reality physical therapy interventions will be assessed using the Feasibility and acceptability survey(patient). Survey contains 10 items. First 5 items are yes no questions. Last 5 items are scored on a Likert scale from 1 to 10 where higher scores indicate higher feasibility.
Feasibility and acceptability survey(parent) | immediately after the physical therapy session
  This is an self developed feasibility survey. Feasibility, of the virtual reality physical therapy interventions will be assessed using the Feasibility and acceptability survey(parent). Survey contains 3 items. Scale items are scored on a Likert scale from 1 to 5 where higher scores indicate higher satisfaction.
Difference in FACIT-F questionnaire result | immediately after the physical therapy session
  Measured by comparison Pediatric Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) of patient in first physical therapy session and second physical therapy session .
  Pediatric Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) is a 13 items -questionnaire which measures the fatigue scale of the patient with minimum score at 0 (low fatigue score) and maximum score at 52 (high fatigue score).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Caruso, Study Director — Stanford University
Locations (1):
- Lucile Packard Childrens Hospital Stanford, Palo Alto, California, United States